CLINICAL TRIAL: NCT05390840
Title: A Phase II Trial to Evaluate the Efficacy and Safety of Topical Ocular MG-O-1002 in Patients With Neovascular Age-Related Macular Degeneration (nAMD)
Brief Title: A Study to Investigate the Effect on Central Macular Thickness of Treatment With MG-O-1002 Eye Drops in Participants Aged Over 45 With Neovascular Age-related Macular Degeneration (nAMD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Theratocular Biotek Co. (Industry)
Responsible Party: Sponsor
Organization: Metagone Biotech Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TO-02C201
Record Dates: First submitted 2022-05-20; First posted 2022-05-25 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-10

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant
Masking Description: Part 1 - Open Label (24 Participants); Part 2 - Single-Blind to Participant (12 Participants)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1 (MG-O-1002) (Experimental): Drug: MG-O-1002; Dose level: 0.8%; Dosage form: ophthalmic solution; Route of administration: topical ocular
  Interventions: Drug: MG-O-1002
- Part 2 (MG-O-1002 or Placebo) (Placebo Comparator): Arm 1:
  Drug: MG-O-1002; Dose level: 0.8%; Dosage form: ophthalmic solution; Route of administration: topical ocular
  Arm 2:
  Drug: Placebo; Dosage form: ophthalmic solution; Route of administration: topical ocular
  Interventions: Drug: MG-O-1002; Other: Placebo

INTERVENTIONS:
Drug: MG-O-1002 — MG-O-1002 ophthalmic solution in one concentration (0.8%) ocular administration 3 drops in study eye
Other: Placebo — The placebo is 0.9% saline ocular administration 3 drops in study eye
  Arms: Part 2 (MG-O-1002 or Placebo)

SUMMARY:
A 2 parts Phase II study to investigate the effect on central macular thickness of treatment with MG-O-1002 eye drops in participants aged over 45 with neovascular age-related macular degeneration (nAMD)

DETAILED DESCRIPTION:
Neovascular Age-related Macular Degeneration (nAMD) is a serious eye disease and a leading cause of irreversible blindness primarily in the older population. Current treatment with anti-vascular endothelial growth factor (VEGF), while effective, requires intravitreal injection meaning administration that needs to be performed by a specialist ophthalmologist and carries procedural risks. MG-O-1002 can be administered as a topical eye drop providing a potentially safer option that can be self-administered increasing accessibility. This study will evaluate the efficacy and safety of topical ocular use of MG-O-1002 in participants with nAMD.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. Adults aged 45 years or older with a diagnosis of nAMD
2. Diagnosis in the study eye of active, pathologic, newly diagnosed and treatment naïve (i.e., no previous anti-VEGF treatment or other surgery in the study eye)
3. Visual acuity from 20/25 to 20/200 in the study eye
4. Total lesion size (including neovascularization, blood) ≦12 disc areas (30.5 mm2) as assessed by Fluorescein Angiography.
5. Demonstrate the ability, or have a family member who is willing and able to, instill topical ocular drops in the study eye.
6. Ability to give written informed consent and comply with study procedures.

Part 2:

1. Adults aged 45 years or older with a diagnosis of nAMD.
2. Participant with nAMD previously treated with 3 injections of Aflibercept within the preceding 4 months, and received the last injection within 30 to 21 days before visit 1 of this study.
3. Demonstrate the ability, or have a family member who is willing and able to, instil topical ocular drops in the study eye.
4. Ability to give written informed consent and comply with study procedures.

Exclusion Criteria:

Part 1:

1. Prior use within the last 2 months, or a high possibility of requiring treatment with anti-VEGF therapy (except the study drug) in both eyes during the study.
2. Abnormal regions identified by Fundus Autofluorescence (FAF) and Optical Coherence Tomography (OCT) involving the center of the fovea are caused by retinal pigment epithelium (RPE) atrophy, RPE tear, photoreceptor attenuation, or fibrosis/scar tissue.
3. Significant retinal serous pigment epithelial detachment (PED) involving the fovea.
4. History of, or current clinical evidence in the study eye of aphakia, diabetic macular edema, any ocular inflammation or infection, pathological myopia, retinal detachment, advanced glaucoma, and/or significant media opacity, including cataract.
5. History or evidence of the following surgeries in the study eye: penetrating keratoplasty or vitrectomy; corneal transplant; corneal or intraocular surgery within 3 months of Screening.
6. Uncontrolled hypertension despite the use of antihypertensive medications.
7. Diagnosis of Type 1 or Type 2 diabetes.
8. Use of medications that in the opinion of the Investigator could interfere with study results.
9. Participation in any investigational drug or device study, systemic or ocular, within the past 3 months.
10. Women who are pregnant or breast feeding.
11. Women of child-bearing potential who are not using an effective form of birth control.
12. Known serious allergies or hypersensitivity to the fluorescein dye used in angiography, or to the components of the MG-O-1002 formulation, or to topical anesthetics.
13. In the opinion of the investigator, subject who is not suitable for or not likely be benefited from the study treatment.

Part 2:

1. More than 30 days between 3rd injection of Aflibercept and Visit 1.
2. Patients who have received 3 injections of Aflibercept within the last 3 months and need continued treatment in the fellow eye.
3. Significant retinal serous pigment epithelial detachment (PED), atrophy, or fibrosis/scar involving the fovea.
4. History or evidence of the following surgeries in the study eye: penetrating keratoplasty or vitrectomy; corneal transplant; corneal or intraocular surgery within 3 months of Screening.
5. Active intraocular inflammation or uveitis or scleritis or episcleritis in the study eye or ocular or periocular infection in either eye.
6. Uncontrolled hypertension despite the use of antihypertensive medications.
7. Diagnosis of Type 1 or Type 2 diabetes.
8. Use of medications that in the opinion of the Investigator could interfere with study results.
9. Participation in any investigational drug or device study, systemic or ocular, within the past 3 months.
10. Women who are pregnant or breast feeding.
11. Women of child-bearing potential who are not using an effective form of birth control.
12. Known serious allergies or hypersensitivity to the fluorescein dye used in angiography, or to the components of the MG-O-1002 formulation, or to topical anesthetics.
13. In the opinion of the investigator, subject who is not suitable for or not likely be benefited from the study treatment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in central macular thickness over 12 weeks. | up to 12 weeks

SECONDARY OUTCOMES:
Mean change from baseline in Best-Corrected Visual Acuity over 12 weeks | up to 12 weeks
Mean Change from baseline in Visual Field over 12 weeks | up to 12 weeks
Mean change from baseline in total area of Choroidal Neovascularization (CNV) over 12 weeks | up to 12 weeks
The number of patients needing rescue treatment within 12 weeks | up to 12 weeks
The time to rescue treatment for needed patients within 12 weeks | up to 12 weeks
Incidence and severity of ocular and systemic adverse events | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Thailand (6):
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Metta Pracharak Hospital, Nakhon Pathom
  - Thammasat University Hospital, Pathum Thani
  - Naresuan University Hospital, Phitsanulok

IPD SHARING:
Plan to Share IPD: No